CLINICAL TRIAL: NCT06880588
Title: Relationship Between Sleep Characteristics and Motor Development and Sensory Processing Skills in Late Premature Infants
Brief Title: Sleep Characteristics in Late Premature Infants
Status: Completed | Type: Observational
Sponsor: Gazi University (Other)
Responsible Party: Principal Investigator, Rabia ZORLULAR, principal investigator, Gazi University
Other Study IDs: late premature and sleep
Record Dates: First submitted 2025-03-14; First posted 2025-03-17 (Actual); Last update posted 2025-06-25 (Actual); Status verified 2025-03

CONDITIONS: Late Preterm Infant; Motor Development; Sleep
Keywords: Sleep; late preterm; motor development; sensory processing skill

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Late preterm: Late preterm infants are defined as infants born between 34 and 36 (+6 days) weeks of gestation. Medical literature places great emphasis on extremely low birth weight and extremely preterm infants, but late preterm infants are also at risk and have mortality rates three times higher than those born full term.
  Interventions: Behavioral: Brief Infant Sleep Questionnaire; Behavioral: Test of Sensory Function in Infants; Behavioral: Peabody Motor Development Scale-2

INTERVENTIONS:
Behavioral: Brief Infant Sleep Questionnaire — The Brief Infant Sleep Questionnaire will be used to assess sleep. Infant sleep problems are among the most common problems presented to healthcare professionals. The extended version of the "Brief Infant Sleep Questionnaire" is a questionnaire developed by Sadeh to assess sleep problems and their causes in early childhood. This questionnaire has been translated into Turkish and assessed sleep environment and sleep problems in infants. It consists of 33 items, is based on parent reports of infant or toddler sleep patterns and is used to validate the data. It is associated with daily records and parent reports of sleep. Its sensitivity in documenting developmental sleep trends is well established
Behavioral: Test of Sensory Function in Infants — It was planned to use the Test of Sensory Function in Infants to evaluate the sensory development of infants. Test of Sensory Function in Infants is frequently used to evaluate the sensory processing
Behavioral: Peabody Motor Development Scale-2 — It was planned to use the Peabody Motor Development Scale-2 to evaluate motor development. The Peabody Motor Development Scale-2 was designed to determine developmental delays in children aged 0-72 months.

SUMMARY:
Studies examining sleep and developmental parameters in infants have primarily focused on either term or extremely preterm infants. However, a review of the existing literature reveals a lack of research investigating sleep characteristics and their relationship with motor and sensory development in late preterm infants. Therefore, the present study aims to evaluate sleep characteristics and explore their association with motor development and sensory processing in late preterm infants, who are at higher risk for developmental delays compared to term infants.

DETAILED DESCRIPTION:
Late preterm infants are defined as those born between 34 and 36 weeks and 6 days of gestational age. Although the medical literature places significant emphasis on extremely low birth weight and extremely preterm infants, late preterm infants are also at risk, with mortality rates three times higher than those of term infants. Born with lungs and brains that are not yet fully matured, late preterm infants may experience complications due to immaturity. Although they often appear healthier and more mature than they are, late preterm infants show significant differences from term infants (born between 37 and 42 weeks of gestation), particularly because their brain development has not yet been completed.

During the final weeks of gestation (34-40 weeks), critical developmental processes occur in the brain, including the formation of synaptic connections, myelination, and the development of cortical folds. Compared to normal term neonates, the late preterm brain appears 20% to 30% smaller, less developed, and less myelinated on magnetic resonance imaging. The sensory system is shaped immediately after birth by both the quantity and type of sensory experiences and continues to develop throughout life. In preterm infants, sensory processing has been associated with immaturity at birth, length of stay in the neonatal intensive care unit, white matter injury, and caregiver education.

Sleep is a critical factor for the healthy development of processes such as brain maturation, motor planning, postural control, and sensory integration, especially during infancy. Sleep is closely linked to brain development and infant behavior, and disruptions in sleep patterns can have profound and long-term effects on an infant's overall health, growth, and well-being in early life. Moreover, sleep plays a crucial role in the formation of persistent neural circuits necessary for early sensory development and the maturation of primary sensory systems in infants. The aim of this study is to investigate the relationship between sleep characteristics and motor development and sensory processing skills in late preterm infants (born between 34 weeks and 36 weeks + 6 days of gestation) who are between 6 and 12 months of corrected age. It is thought that sleep problems, which are frequently observed in preterm infants, may have significant effects on motor and sensory development. In this context, the primary objective of the study is to elucidate how sleep patterns and characteristics are associated with motor and sensory development in late preterm infants, and to provide scientific evidence to inform early intervention programs.

ELIGIBILITY:
Inclusion Criteria:

* Late preterm infants with a corrected age of 6-12 months,
* Infants with parental consent

Exclusion Criteria:

* Infants with chromosomal abnormalities,
* having serious congenital problems,
* whose parents are unwilling to work,

Ages: 6 Months to 12 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: The study group will consist of late premature babies (34-36 weeks) and their families whose corrected gestational age is between 6-12 months and whose parents' consent has been obtained.
Sampling Method: Non-Probability Sample
Enrollment: 81 (Actual)
Dates: Start 2025-03-19 (Actual); Primary Completion 2025-06-01 (Actual); Study Completion 2025-06-01 (Actual)

PRIMARY OUTCOMES:
Peabody Developmental Motor Scales | Second Edition | 6-12 months
  It is planned to use Peabody Motor Development Scale-2 to evaluate motor development. The test is designed to determine developmental delays in children between 0-72 months. It is used to evaluate the motor development of children with separate tests and rating scales for both gross motor skills and fine motor skills. Six subtests, reflexes, Stationary, Locomotion, Object Manipulation, Grasping, and Visual-Motor Integration, collectively measure a broad spectrum of motor functions including postural control, locomotor abilities, object manipulation, and hand-eye coordination. The subtests generate three composite scores: the Gross Motor Quotient, Fine Motor Quotient, and Total Motor Quotient, offering a comprehensive evaluation of a child's motor competence. Notably, higher scores on the Peabody Motor Development Scale-2 reflect superior motor performance, indicating better developmental outcomes.
Test of Sensory Functions in Infants | 6-12 months
  It is used to determine whether a infant has a sensory processing problem and to what extent. It consists of 24 items. Test of sensory function in infants requires the baby to be stimulated and interacted with various materials. The total score varies between 0-49 and the test has norm values for different age groups. Although it is used from the fourth month onwards, the most reliable and valid results are obtained between 7-18 months.
Brief Infant Sleep Questionnaire | 6-12 months
  The Brief Infant Sleep Questionnaire will be used to assess sleep. Infant sleep problems are among the most common problems presented to pediatricians. The extended version of the "Brief Infant Sleep Questionnaire" is a questionnaire developed by Sadeh to assess sleep problems and their causes in early childhood. Consists of 33 items, based on parent reports of infant or toddler sleep patterns, and used to validate data. Correlated with daily records and parent reports of sleep. Well-established for accuracy in documenting developmental sleep trends. In scoring, it is categorized as sleep duration, wakefulness duration, number of awakenings from sleep, presence of snoring, location of sleep.

CONTACTS AND LOCATIONS:
Overall Officials: Rabia ZORLULAR, Principal Investigator — Gazi University
Locations (1):
- Gazi University, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Sadeh A, Mindell JA, Luedtke K, Wiegand B. Sleep and sleep ecology in the first 3 years: a web-based study. J Sleep Res. 2009 Mar;18(1):60-73. doi: 10.1111/j.1365-2869.2008.00699.x. Epub 2008 Oct 16. PMID 19021850
- [Background] DeGangi GA, Greenspan SI. The development of sensory functions in infants. Physical & Occupational Therapy in Pediatrics. 1989;8(4):21-33.
- [Background] Young PC, Glasgow TS, Li X, Guest-Warnick G, Stoddard G. Mortality of late-preterm (near-term) newborns in Utah. Pediatrics. 2007 Mar;119(3):e659-65. doi: 10.1542/peds.2006-2486. PMID 17332185
- [Background] Medoff-Cooper B, Bakewell-Sachs S, Buus-Frank ME, Santa-Donato A; Near-Term Infant Advisory Panel. The AWHONN Near-Term Infant Initiative: a conceptual framework for optimizing health for near-term infants. J Obstet Gynecol Neonatal Nurs. 2005 Nov-Dec;34(6):666-71. doi: 10.1177/0884217505281873. PMID 16282223
- [Derived] Zorlular R, Zorlular A, Elbasan B. Relationship between sleep characteristics, motor development, and sensory processing in late preterm infants. Sleep Med. 2025 Dec;136:106851. doi: 10.1016/j.sleep.2025.106851. Epub 2025 Oct 13. PMID 41106044